CLINICAL TRIAL: NCT03428399
Title: Risk and Protective Factors for Depression and Body Image Distress Following Mastectomy With Breast Reconstruction
Brief Title: Depression and Body Image Distress Following Mastectomy With Reconstruction
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Hilary Weingarden, Psychologist, Massachusetts General Hospital
Other Study IDs: 2017P000944
Record Dates: First submitted 2018-02-05; First posted 2018-02-09 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer; BRCA1 Mutation; BRCA2 Mutation
Keywords: breast reconstruction; mastectomy
MeSH Terms: conditions — Breast Neoplasms | interventions — Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast reconstruction patients: Self-reported psychosocial variables and a clinical interview assessing mental health history will be administered prior to participants' scheduled mastectomy and breast reconstruction surgery (which is part of their routine medical care for cancer treatment or prevention). Follow up self-report measures will be collected after the surgery as well.
  Interventions: Other: Psychosocial variables

INTERVENTIONS:
Other: Psychosocial variables — The investigators will assess mental health history and self-reported psychosocial variables as hypothesized risk and protective factors for body image and depression severity in breast reconstruction patients, before and after their mastectomy and breast reconstruction surgery. Mastectomy and breast reconstruction will be received in the context of routine medical care. Thus, this is not a psychological intervention, but rather observational measures assessed pre- and post routine care for breast reconstruction patients.

SUMMARY:
Mastectomy is a major surgery that can have a profound effect on women's psychosocial wellbeing, including elevated depression and body image distress. Reconstructive breast surgery aims to improve patients' psychosocial adjustment to mastectomy, yet for some women substantial distress persists after reconstruction. However, very little is known about risk or protective factors for persistent depression or body image distress following mastectomy with reconstruction. The present study aims to address this critical gap. In women undergoing mastectomy with breast reconstruction, the investigators will assess risk and protective factors for post-surgery depression severity and body image distress.

ELIGIBILITY:
Inclusion Criteria:

1. Female adults (age 18+) who are scheduled for mastectomy with immediate breast reconstruction at the Massachusetts General Hospital (MGH) Plastic and Reconstructive Surgery Program
2. English language proficiency
3. Ability to provide informed consent.

Exclusion Criteria:

1. Current psychotic disorder, manic episode, serious neurological disorder, intellectual disability, or developmental disorder
2. Current active suicidal ideation
3. Current treatment plan includes radiation and/or ongoing chemotherapy
4. Does not have access to Internet at home, required to complete study questionnaires

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who are scheduled for mastectomy with immediate breast reconstruction at Massachusetts General Hospital as part of their routine medical care. The treatment plan for eligible participants may not include chemotherapy or radiation at the time of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-05-03 (Actual)

PRIMARY OUTCOMES:
Body Image Scale (BIS) | 2-3 months post-surgery (i.e., Time 2)
  Assesses severity of body image distress related to breast cancer treatment with a summed total score, which ranges from 0 (no body image distress) to 30 (substantial body image distress).
Beck Depression Inventory-II (BDI-II) | 2-3 months post-surgery (i.e., Time 2)
  Assesses severity of depressive symptoms with a summed total score, which ranges from 0 (no depressive symptoms) to 63 (severe depressive symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Hilary Weingarden, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weingarden H, Laky ZE, Ladis I, Austen WG Jr, Wilhelm S. Body Image After Mastectomy Scale: A New Measure of Body Image Behaviors and Beliefs in Women Following Mastectomy. J Womens Health (Larchmt). 2022 Jan;31(1):47-54. doi: 10.1089/jwh.2021.0131. Epub 2021 Aug 26. PMID 34449252